CLINICAL TRIAL: NCT05682833
Title: Adjunctive Use Of A Novel Hyaluronic Acid/Chlorhexidine Gel In The Non Surgical Treatment Of Periodontitis: A Split Mouth Randomized Controlled Trial
Brief Title: Adjunctive Use Of A Novel Hyaluronic Acid/Chlorhexidine Gel In The Non Surgical Treatment Of Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Zahi BADRAN, Professor, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-22-02-26-S
Record Dates: First submitted 2022-12-28; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Periodontitis; Hyaluronic Acid; Chlorhexidine
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Split mouth RCT
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): NS therapy + Chlorhexidine/Hyaluronic acid subgingival gel application
  Interventions: Procedure: Non surgical periodontal therapy
- Control (Placebo Comparator): NS therapy + Placebo gel subgingival application
  Interventions: Procedure: Non surgical periodontal therapy

INTERVENTIONS:
Procedure: Non surgical periodontal therapy — Subgingival ultrasonic debridement + manual root planning

SUMMARY:
General Objective :

To evaluate the outcome of non surgical periodontal therapy with local drug delivery adjunct to scaling and root planning

Specific Objective :

To determine the effect of intra-pocket application of hyaluronic acid /chlorohexidine gel in non surgical periodontal treatment on clinical periodontal parameters and microbiological level .

ELIGIBILITY:
Inclusion Criteria:

* Age : 20-60 years old
* At least 20 remaining teeth
* Periodontitis stage III and IV ,Grade A, B and C

Exclusion Criteria:

* Patients taking specific medications: antibiotic , anticoagulants or anti-inflammatory
* Previous periodontal therapy in the past 3-6 months.
* Immunocompromised patients
* Systemically diseased patients: Diabetes ,osteoporosis etc
* History of allergies or hypersensitivity reactions to chlorohexidine or Hyaluronic acid
* Pregnant or lactating women.
* Heavy Smokers (more than 20/day)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
pocket depth | 2 months
Bleeding on Probing | 2 months
Clinical attachment level | 2 months

SECONDARY OUTCOMES:
Plaque index | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Zahi BADRAN, Phd, Study Director — University of Sharjah
Locations (1):
- University Dental Hospital Sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No